CLINICAL TRIAL: NCT02431247
Title: A Phase 3, Randomized, Active-controlled, Double-blind Study to Evaluate Efficacy and Safety of Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (D/C/F/TAF) Once Daily Fixed Dose Combination Regimen Versus a Regimen Consisting of Darunavir/Cobicistat Fixed Dose Combination Coadministered With Emtricitabine/Tenofovir Disoproxil Fumarate Fixed Dose Combination in Antiretroviral Treatment-naive Human Immunodeficiency Virus Type 1 Infected Subjects
Brief Title: A Study to Evaluate Efficacy and Safety of Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (D/C/F/TAF) Fixed Dose Combination (FDC) Versus a Regimen Consisting of Darunavir/Cobicistat FDC With Emtricitabine/Tenofovir Disoproxil Fumarate FDC in Treatment-naive HIV Type 1 Infected Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR107277; TMC114FD2HTX3001 (Other: Janssen Sciences Ireland UC); 2015-000754-38 (EudraCT Number)
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Immunodeficiency Virus Type 1, Human
Keywords: Immunodeficiency Virus Type 1, Human; Darunavir; Cobicistat; Tenofovir Alafenamide; Emtricitabine; Tenofovir Disoproxil Fumarate
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Darunavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (Experimental): Subject will receive a single oral tablet containing darunavir (DRV) 800 milligram (mg)/ cobicistat (COBI) 150 mg/ emtricitabine (FTC) 200 mg/ tenofovir alafenamide (TAF) 10 mg (D/C/F/TAF fixed dose combination [FDC]) once daily along with DRV/COBI FDC-matching and FTC/TDF FDC-matching placebo tablets once daily up to Week 48 analysis unblinding visit (i.e. after last subject has reached Week 48). After Week 48 analysis unblinding visit, subjects will receive a single tablet containing D/C/F/TAF FDC once daily up to Week 96.
  Interventions: Drug: Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide FDC; Drug: FTC/TDF FDC Matching Placebo; Drug: DRV/COBI FDC Matching Placebo
- DRV/COBI fixed dose combination (FDC) and FTC/TDF FDC (Active Comparator): Subject will receive DRV 800 mg/COBI 150 mg FDC and FTC 200 mg/TDF 300 mg FDC along with D/C/F/TAF FDC-matching placebo tablet once daily up to Week 48 analysis unblinding (i.e. after last subject has reached Week 48). After Week 48 analysis unblinding, subjects will receive a single tablet containing D/C/F/TAF FDC once daily up to Week 96.
  Interventions: Drug: DRV/COBI FDC; Drug: FTC/TDF FDC; Drug: D/C/F/TAF FDC - Matching Placebo

INTERVENTIONS:
Drug: Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide FDC — A tablet containing DRV 800 mg, COBI 150 mg, FTC 200 mg and TAF) 10 mg will be administered once daily.
  Arms: Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide
Drug: DRV/COBI FDC — A tablet containing DRV 800 mg and COBI 150 mg will be administered once daily.
  Arms: DRV/COBI fixed dose combination (FDC) and FTC/TDF FDC
Drug: FTC/TDF FDC — A tablet containing FTC 200 mg and TDF 300 mg will be administered once daily.
  Arms: DRV/COBI fixed dose combination (FDC) and FTC/TDF FDC
Drug: D/C/F/TAF FDC - Matching Placebo — Matching placebo of D/C/F/TAF FDC will be administered once daily.
  Arms: DRV/COBI fixed dose combination (FDC) and FTC/TDF FDC
Drug: FTC/TDF FDC Matching Placebo — Matching placebo of FTC/TDF FDC will be administered once daily.
  Arms: Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide
Drug: DRV/COBI FDC Matching Placebo — Matching placebo of DRV/COBI FDC will be administered once daily.
  Arms: Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide

SUMMARY:
The purpose of this study is to demonstrate non-inferiority in efficacy of a darunavir/cobicistat/emtricitabine/tenofovir alafenamide (D/C/F/TAF) fixed dose combination (FDC) tablet versus Darunavir/Cobicistat (DRV/COBI) FDC coadministered with Emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) FDC in human immunodeficiency virus-1 (HIV-1) infected, antiretroviral (ARV) treatment naive adult participants.

DETAILED DESCRIPTION:
This is a Phase 3, multicenter (when more than one hospital or medical school team work on a medical research study), randomized (study drug assigned by chance), double-blind (a medical research study in which neither the researchers nor the participant know what treatment the participant is receiving), active-controlled (study in which the experimental treatment or procedure is compared to a standard [control] treatment or procedure) study. The study consists of 5 periods: a Screening period, Double-blind treatment period, Single-arm treatment period, Extension period and a Follow-up period. Participants will receive either darunavir (DRV)/ cobicistat (COBI)/emtricitabine (FTC) /tenofovir alafenamide (TAF) fixed dose combination (D/C/F/TAF FDC) or DRV/COBI FDC along with FTC/TDF FDC. Primarily percentage of participants with human immunodeficiency virus (HIV) -1 Ribonucleic acid (RNA) less than (<) 50 copies per milliliter (copies/ml) defined by snapshot analysis will be evaluated. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be antiretroviral (ARV) treatment-naive (never treated with an ARV including post-exposure prophylaxis and pre-exposure prophylaxis); no prior use of any approved or experimental anti- human immunodeficiency virus (anti-HIV) drug for any length of time
* Screening plasma HIV-1 ribonucleic acid (RNA) level greater than or equal to >=1,000 copies per milliliter (copies/mL)
* Cluster of Differentiation 4+ (CD4+) cell count >50 cells/microliter (cells/mcL)
* Screening HIV-1 genotype report must show full sensitivity to DRV, TDF and FTC
* Screening eGFRcreatinine >=70 mL/min according to the Cockcroft-Gault formula for creatinine clearance

Exclusion Criteria:

* Subject has been diagnosed with a new acquired immunodeficiency syndrome (AIDS)-defining condition within the 30 days prior to screening
* Subject has proven or suspected acute hepatitis within 30 days prior to screening
* Subject is hepatitis C or hepatitis B positive
* Subject has a history of cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 725 (Actual)
Dates: Start 2015-07-06 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (80):
- United States (29):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Bakersfield, California
  - Long Beach, California
  - Los Angeles, California
  - North Hollywood, California
  - San Francisco, California
  - Washington D.C., District of Columbia
  - Ft. Pierce, Florida
  - Miami, Florida
  - Orlando, Florida
  - West Palm Beach, Florida
  - Savannah, Georgia
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Berkley, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Hillsborough, New Jersey
  - Newark, New Jersey
  - Somers Point, New Jersey
  - Santa Fe, New Mexico
  - Manhasset, New York
  - Chapel Hill, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Fort Worth, Texas
  - Houston, Texas
  - Seattle, Washington
- Belgium (3):
  - Antwerp
  - Brussels
  - Ghent
- Canada (2):
  - Toronto, Ontario
  - Montreal, Quebec
- France (9):
  - Clamart
  - Le Kremlin-Bicêtre
  - Lyon
  - Marseille
  - Montpellier
  - Nantes
  - Paris
  - Strasbourg
  - Tourcoing
- Germany (9):
  - Berlin
  - Bonn
  - Cologne
  - Essen
  - Frankfurt
  - Freiburg im Breisgau
  - Hamburg
  - Hanover
  - München
- Poland (7):
  - Bydgoszcz
  - Chorzów
  - Krakow
  - Lodz
  - Szczecin
  - Warsaw
  - Wroclaw
- San Juan, Puerto Rico
- Russia (8):
  - Krasnodar
  - Oryol
  - Saint Petersburg
  - Saratov
  - Smolensk
  - Tolyatti
  - Voronezh
  - Yekaterinburg
- Spain (9):
  - Alicante
  - Badalona
  - Barcelona
  - Córdoba
  - Elche
  - Madrid
  - Santiago de Compostela
  - Seville
  - Valencia
- United Kingdom (3):
  - Brighton
  - Bristol
  - London

REFERENCES:
- [Derived] Ackaert O, McDougall D, Perez-Ruixo C, Perez-Ruixo JJ, Jezorwski J, Crauwels HM. Population Pharmacokinetic Analysis of Darunavir and Tenofovir Alafenamide in HIV-1-Infected Patients on the Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide Single-Tablet Regimen (AMBER and EMERALD Studies). AAPS J. 2021 Jun 7;23(4):82. doi: 10.1208/s12248-021-00607-8. PMID 34100149
- [Derived] Orkin C, Eron JJ, Rockstroh J, Podzamczer D, Esser S, Vandekerckhove L, Van Landuyt E, Lathouwers E, Hufkens V, Jezorwski J, Opsomer M; AMBER study group. Week 96 results of a phase 3 trial of darunavir/cobicistat/emtricitabine/tenofovir alafenamide in treatment-naive HIV-1 patients. AIDS. 2020 Apr 1;34(5):707-718. doi: 10.1097/QAD.0000000000002463. PMID 31833849
- [Derived] Lathouwers E, Wong EY, Brown K, Baugh B, Ghys A, Jezorwski J, Mohsine EG, Van Landuyt E, Opsomer M, De Meyer S; AMBER and EMERALD Study Groups. Week 48 Resistance Analyses of the Once-Daily, Single-Tablet Regimen Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (D/C/F/TAF) in Adults Living with HIV-1 from the Phase III Randomized AMBER and EMERALD Trials. AIDS Res Hum Retroviruses. 2020 Jan;36(1):48-57. doi: 10.1089/AID.2019.0111. Epub 2019 Oct 21. PMID 31516033
- [Derived] Rashbaum B, Spinner CD, McDonald C, Mussini C, Jezorwski J, Luo D, Van Landuyt E, Brown K, Wong EY. Darunavir/cobicistat/emtricitabine/tenofovir alafenamide in treatment-naive patients with HIV-1: subgroup analyses of the phase 3 AMBER study. HIV Res Clin Pract. 2019 Feb;20(1):24-33. doi: 10.1080/15284336.2019.1608714. Epub 2019 May 29. PMID 31303147
- [Derived] Eron JJ, Orkin C, Gallant J, Molina JM, Negredo E, Antinori A, Mills A, Reynes J, Van Landuyt E, Lathouwers E, Hufkens V, Jezorwski J, Vanveggel S, Opsomer M; AMBER study group. A week-48 randomized phase-3 trial of darunavir/cobicistat/emtricitabine/tenofovir alafenamide in treatment-naive HIV-1 patients. AIDS. 2018 Jul 17;32(11):1431-1442. doi: 10.1097/QAD.0000000000001817. PMID 29683855

RESULTS

PARTICIPANT FLOW:
Groups:
- D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]): Participants received a single oral tablet containing darunavir (DRV) 800 milligram (mg)/ cobicistat (COBI) 150 mg/ emtricitabine (FTC) 200 mg/ tenofovir alafenamide (TAF) 10 mg (D/C/F/TAF fixed dose combination [FDC]) once daily along with DRV/COBI FDC-matching placebo and FTC/tenofovir disoproxil fumarate (TDF) FDC-matching placebo tablets once daily up to Week 48 analysis unblinding visit (that is, after last participant has reached Week 48). After Week 48 analysis unblinding visit, all participants received D/C/F/TAF treatment up to Week 96 during the open-label, single-group treatment phase. After Week 96, participants were given the opportunity to continue D/C/F/TAF treatment during an extension phase until the D/C/F/TAF FDC tablet became commercially available.
- DRV/COBI+ FTC/TDF (Control) (Baseline to Switch): Participants received DRV 800 mg/COBI 150 mg FDC and FTC 200 mg/TDF 300 mg FDC along with D/C/F/TAF FDC-matching placebo tablet once daily Subjects received DRV 800 mg/COBI 150 mg FDC and FTC 200 mg/TDF 300 mg FDC along with D/C/F/TAF FDC-matching placebo tablet once daily up to Week 48 analysis unblinding visit (that is, after last subject has reached Week 48).
- Switch to D/C/F/TAF: After Week 48 analysis unblinding visit, participants earlier receiving treatment with DRV/COBI+ FTC/TDF (Control) switched to D/C/F/TAF treatment and continued for up to Week 96 during open-label, single-group treatment phase. After Week 96, participants were given the opportunity to continue D/C/F/TAF treatment until the D/C/F/TAF FDC tablet became commercially available.
Period: BL to EOE-Test and BL to Switch- Control
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch) | Switch to D/C/F/TAF
Started | 362 | 363 | 0
Completed | 296 | 322 | 0
Not Completed | 66 | 41 | 0
Not completed — Other | 11 | 2 | 0
Not completed — Lost to Follow-up | 17 | 8 | 0
Not completed — Physician Decision | 9 | 4 | 0
Not completed — Pregnancy | 1 | 1 | 0
Not completed — Adverse Event | 12 | 16 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Withdrawal by Subject | 14 | 9 | 0
Not completed — Subject non-compliant | 2 | 0 | 0
Period: Switch to D/C/F/TAF (Until EOE)
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch) | Switch to D/C/F/TAF
Started | 0 | 0 (322 participants from DRV/COBI+ FTC/TDF (Control) group switched to D/C/F/TAF (Test) Group) | 322 (322 participants from DRV/COBI+ FTC/TDF (Control) group switched to D/C/F/TAF (Test) Group)
Completed | 0 | 0 | 289
Not Completed | 0 | 0 | 33
Not completed — Other | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 12
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 5
Not completed — Death | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 10

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included all the participants who were randomized and received at least one dose of study treatment in the study.
Groups:
- D/C/F/TAF (Test) (Baseline to End of Extension [EOE]): Participants received a single oral tablet containing darunavir (DRV) 800 milligram (mg)/ cobicistat (COBI) 150 mg/ emtricitabine (FTC) 200 mg/ tenofovir alafenamide (TAF) 10 mg (D/C/F/TAF fixed dose combination [FDC]) once daily along with DRV/COBI FDC-matching placebo and FTC/tenofovir disoproxil fumarate (TDF) FDC-matching placebo tablets once daily up to Week 48 analysis unblinding visit (that is, after last participant has reached Week 48). After Week 48 analysis unblinding visit, all participants received D/C/F/TAF treatment up to Week 96 during the open-label, single-group treatment phase. After Week 96, participants were given the opportunity to continue D/C/F/TAF treatment during an extension phase until the D/C/F/TAF FDC tablet became commercially available.
- Total: Total of all reporting groups
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch) | Total
Number analyzed (Participants) | 362 | 363 | 725
Age, Continuous [Median (Full Range); unit: years] | 34 [19 to 61] | 34 [18 to 71] | 34.0 [18 to 71]
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0
  Adults (18-64 years) | 362 | 362 | 724
  From 65 to 84 years | 0 | 1 | 1
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 41 | 85
  Male | 318 | 322 | 640
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 7 | 11
  Black or African American | 40 | 40 | 80
  Hispanic or Latino | 41 | 38 | 79
  Other | 19 | 18 | 37
  White Non-Hispanic | 258 | 260 | 518

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Human Immunodeficiency Virus (HIV)-1 Ribonucleic Acid (RNA) Less Than (<) 50 Copies Per Milliliter (Copies Per mL) (Virologic Response) at Week 48 Defined by Food and Drug Administration (FDA) Snapshot Approach
Description: Percentage of participants with a HIV-1 RNA < 50 copies per mL were assessed using FDA snapshot approach which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status. The snapshot approach classified participants into 3 outcome categories: 1) virologic success (HIV RNA < 20/50/200 copies per mL at Week 48), 2) virologic failure (HIV RNA greater than or equal to [>=] 20/50/200 copies per mL at Week 48), 3) no viral load data in the Week 48 visit window (discontinued due to adverse event/death/other reason). The missing HIV-1 RNA is considered as non-response.
Time Frame: At Week 48
Population: The intent-to-treat (ITT) analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Here N (number of participants analyzed) refers to 362 for test group and 363 for control group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch)
Number analyzed (Participants) | 362 | 363
percentage of participants | 91.4 (88.1) [88.1 to 94.1] | 88.4 (84.7) [84.7 to 91.5]
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) vs DRV/COBI+ FTC/TDF (Control) (Baseline to Switch); Test type: Non-Inferiority — One-sided p-value for non-inferiority of Test versus Control arm. The non-; p < 0.001, Mantel Haenszel — inferiority margin is 10%; Difference in percentage = 2.7, 95% CI 2-sided [-1.6 to 7.1]

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA <20 and 200 Copies Per mL at Weeks 48 and 96 Defined by FDA Snapshot Approach
Description: Percentage of participants with HIV-1 RNA < 20/200 copies per mL using FDA snapshot approach were reported. The snapshot approach classified participants into 3 outcome categories: 1) virologic success (HIV RNA < 20/50/200 copies per mL at Week 48 and 96), 2) virologic failure (HIV RNA >= 20/50/200 copies per mL at Week 48 and 96), 3) no viral load data in the Week 48 and 96 visit window (discontinued due to adverse event/death/other reason). The missing HIV-1 RNA is considered as non-response.
Time Frame: At Weeks 48 and 96
Population: The analysis population is ITT. Here, N (number of participants analyzed) signifies participants evaluated for this outcome measure and n (number analyzed) signifies participants analyzed for this OM for specific categories at specified timepoints. Participants received treatment from baseline till Week 48/Switch in control arm and from switch till Week 96 in Switch to D/C/F/TAF arm. Therefore, Week 96 and Week 48 data was not collected for both arms at respective timepoints.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch) | Switch to D/C/F/TAF
Number analyzed (Participants) | 362 | 363 | 291
percentage of participants
  At week 48: <20 Copies per mL: number analyzed (Participants) | 362 | 363 | 0
  At week 48: <20 Copies per mL | 82.6 [78.3 to 86.4] | 79.3 [74.8 to 83.4] |
  At week 48: <200 Copies per mL: number analyzed (Participants) | 362 | 363 | 0
  At week 48: <200 Copies per mL | 92.8 [89.7 to 95.3] | 90.6 [87.2 to 93.4] |
  At week 96: <20 Copies per mL: number analyzed (Participants) | 362 | 0 | 291
  At week 96: <20 Copies per mL | 76.2 [71.5 to 80.5] |  | 83.5 [78.7 to 87.6]
  At week 96: <200 Copies per mL: number analyzed (Participants) | 362 | 0 | 291
  At week 96: <200 Copies per mL | 86.2 [82.2 to 89.6] |  | 96.9 [94.2 to 98.6]

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 20, 50, and 200 Copies Per mL at Week 48 and 96 Defined by the Time to Loss of Virologic Response (TLOVR) Algorithm
Description: Percentage of participants with HIV-1 RNA less than (<) 20, 50, and 200 copies per mL at Weeks 48 and 96 based on TLOVR algorithm were assessed. TLOVR requires sustained HIV-1 RNA < 50 copies per mL; confirmed HIV-1 RNA >= 50 copies per mL is considered as non-response (rebound); participant is considered non-responder after permanent discontinuation.
Time Frame: At Week 48 and 96
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch) | Switch to D/C/F/TAF
Number analyzed (Participants) | 362 | 363 | 291
percentage of participants
  At Week 48: < 20 Copies per mL: number analyzed (Participants) | 362 | 363 | 0
  At Week 48: < 20 Copies per mL | 82.6 [78.3 to 86.4] | 79.9 [75.4 to 83.9] |
  At Week 48: <50 Copies per mL: number analyzed (Participants) | 362 | 363 | 0
  At Week 48: <50 Copies per mL | 91.2 [87.8 to 93.9] | 88.7 [85.0 to 91.8] |
  At Week 48: <200 Copies per mL: number analyzed (Participants) | 362 | 363 | 0
  At Week 48: <200 Copies per mL | 93.1 [90.0 to 95.5] | 91.7 [88.4 to 94.4] |
  At Week 96: <20 Copies per mL: number analyzed (Participants) | 362 | 0 | 291
  At Week 96: <20 Copies per mL | 73.2 [68.3 to 77.7] |  | 78.4 [73.2 to 82.9]
  At Week 96: <50 Copies per mL: number analyzed (Participants) | 362 | 0 | 291
  At Week 96: <50 Copies per mL | 85.1 [81.0 to 88.6] |  | 93.8 [90.4 to 96.3]
  At Week 96: <200 Copies per mL: number analyzed (Participants) | 362 | 0 | 291
  At Week 96: <200 Copies per mL | 86.7 [82.8 to 90.1] |  | 96.9 [94.2 to 98.6]

4. Secondary Outcome: Change From Baseline in log10 HIV-1 RNA Levels at Week 48
Description: Change from baseline in log10 HIV-1 RNA levels were reported.
Time Frame: Baseline and Week 48
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Based on not completed (NC) equal to (=) failure (F) analysis with values after discontinuation imputed with the baseline value. Other (intermittent) missing values are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: log10 HIV-1 RNA copies per mL
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch)
Number analyzed (Participants) | 362 | 363
log10 HIV-1 RNA copies per mL | -2.95 (0.044) [lower limit 0.044] | -2.91 (0.044) [lower limit 0.044]
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) vs DRV/COBI+ FTC/TDF (Control) (Baseline to Switch); Test type: Other; p = 0.437, ANCOVA; Least square mean difference = -0.05, 95% CI 2-sided [-0.171 to 0.074], Standard Error of Mean 0.063

5. Secondary Outcome: Change From Baseline in Cluster of Differentiation-4 (CD4+) Cell Count at Week 48
Description: The immunologic change was determined by changes in Cluster of CD4+ cell count. Change from baseline in CD4+ cell count at Week 48 were assessed.
Time Frame: Baseline and Week 48
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Based on NC = F analysis with values after discontinuation imputed with the baseline value. Other (intermittent) missing values are imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: Cells per millimeter cube (cells/mm^3)
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch)
Number analyzed (Participants) | 362 | 363
Cells per millimeter cube (cells/mm^3) | 190.49 (10.472) [lower limit 10.472] | 172.01 (10.458) [lower limit 10.458]
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) vs DRV/COBI+ FTC/TDF (Control) (Baseline to Switch); Test type: Other; p = 0.213, ANCOVA; LS mean difference = 18.48, 95% CI 2-sided [-10.595 to 47.550], Standard Error of Mean 14.808

6. Secondary Outcome: Change From Baseline in Serum Creatinine at Week 48
Description: Change from baseline in serum creatinine at Week 48 was reported.
Time Frame: Baseline and Week 48
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Here, N (number of participants analyzed) signifies participants evaluated for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: milligram per deciliter (mg/dL)
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch)
Number analyzed (Participants) | 340 | 330
milligram per deciliter (mg/dL) | 0.05 (0.006) [lower limit 0.006] | 0.09 (0.006) [lower limit 0.006]
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) vs DRV/COBI+ FTC/TDF (Control) (Baseline to Switch); Test type: Other; p < 0.001, ANCOVA; LS mean difference = -0.04, 95% CI 2-sided [-0.05 to -0.02], Standard Error of Mean 0.008

7. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate Based on Serum Creatinine (eGFRcr) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Formula at Week 48
Description: Change from baseline in eGFRcr was calculated using the CKD-EPI equation as per which Stage 1 (normal or high GFR [>=90 mL/min]); Stage 2 (Mild CKD [60 to 90 mL/min]); Stage 3 (Moderate CKD [30 to 59mL/min]); Stage 4 (Severe CKD [15 to 29 mL/min]); Stage 5 (End Stage CKD [<15 mL/min]). The eGFRcr was assessed by calculating serum creatinine (Scr) using the equation: eGFRcr milliliter per minute per 1.72 meter square (mL/min/1.73m^2) = 144*(Scr/0.7)^-0.329*0.993^age (Scr =< 0.7 mg/dL) and eGFRcr mL/min/1.73m^2 = 144*(Scr/0.7)^-1.209*0.993^age (Scr >0.7 mg/dL) for female participants and eGFRcr mL/min/1.73m^2 = 141*(Scr/0.9)^-0.411*0.993^age (Scr =<0.9 mg/dL) and eGFRcr mL/min/1.73m^2 = 141*(Scr/0.9)^-1.209*0.993^age (Scr >0.9 mg/dL) for male participants.
Time Frame: Baseline and Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch)
Number analyzed (Participants) | 340 | 330
mL/min/1.73 m^2 | -6.04 (0.551) [lower limit 0.551] | -9.16 (0.559) [lower limit 0.559]
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) vs DRV/COBI+ FTC/TDF (Control) (Baseline to Switch); Test type: Other; p < 0.001, ANCOVA; LS mean difference = 3.12, 95% CI 2-sided [1.57 to 4.66], Standard Error of Mean 0.786

8. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate Based on Serum Creatinine by (Cockcroft-Gault Formula) at Week 48
Description: Change from baseline in eGFRcr by cockcroft-gault formula at Week 48. The eGFRcr was assessed by calculated creatinine clearance (CrCl) using the Cockcroft-Gault formula, and was assessed using CrCl [mL/min] = (140 - A) * W / (72 * C) * R. Where A is age at sample date [years], W is body weight at specific visit (kilogram [kg]), C is the serum concentration of creatinine [mg/dL], R = 1 if the participant is male and = 0.85 if female.
Time Frame: Baseline and Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: milliliter per minute (mL/min)
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch)
Number analyzed (Participants) | 340 | 330
milliliter per minute (mL/min) | -5.16 (0.790) [lower limit 0.790] | -11.20 (0.802) [lower limit 0.802]
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) vs DRV/COBI+ FTC/TDF (Control) (Baseline to Switch); Test type: Other; p < 0.001, ANCOVA; LS mean difference = 6.04, 95% CI 2-sided [3.83 to 8.25], Standard Error of Mean 1.126

9. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate Based on Serum Cystatin C (eGFRcyst) by CKD-EPI Formula at Week 48
Description: Change from baseline in eGFRcyst was calculated using the CKD-EPI equation as per which Stage 1 (normal or high GFR) >= 90 indicates normal kidney function; Stage 2 (Mild CKD): 60 to 89 mL/min indicates mildly reduced kidney function; Stage 3 (Moderate CKD): 30 to 59 mL/min indicates moderately reduced kidney function; Stage 4 (Severe CKD): 15 to 29 mL/min indicates severely reduced kidney function; Stage 5 (End Stage of CKD): <15 mL/min indicate very severe or end stage kidney failure. The eGFRcyst was assessed by calculated serum cystatin C (Scyst) using the equation: eGFRcyst mL/min/1.73m^2 = 133 * (Scyst/0,8)^-0.499 * 0.996^age [* 0.932 if female] (Scyst =<0.8 mg/L) and eGFRcr mL/min/1.73m^2 = 133 * (Scyst/0,8)^-1.328 * 0.996^age [* 0.932 if male] (Scyst >0.8 mg/L).
Time Frame: Baseline and Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch)
Number analyzed (Participants) | 337 | 329
mL/min/1.73 m^2 | 5.32 (0.525) [lower limit 0.525] | 2.92 (0.532) [lower limit 0.532]
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) vs DRV/COBI+ FTC/TDF (Control) (Baseline to Switch); Test type: Other; p = 0.001, ANCOVA; LS mean difference = 2.40, 95% CI 2-sided [0.93 to 3.87], Standard Error of Mean 0.747

10. Secondary Outcome: Percentage of Participants With Grade 3 and 4 Adverse Events (AEs), Serious Adverse Events (SAEs), and Premature Discontinuations Due to Adverse Events Through Week 48
Description: AE is any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Events with Grade 3 or higher (3=Severe; 4=life-threatening; 5=fatal) are events that significantly interrupt usual daily activity, require systemic drug therapy/other treatment and are, in many situations, considered unacceptable or intolerable events. SAE is any adverse event (AE) that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Up to Weeks 48
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study.
Measure: Number; unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch)
Number analyzed (Participants) | 362 | 363
percentage of participants
  Grade 3 AEs | 4.7 | 4.4
  Grade 4 AEs | 0.6 | 1.7
  SAEs | 4.7 | 5.8
  Premature discontinuations due to AEs | 1.9 | 4.4

11. Secondary Outcome: Change From Baseline in Urine Protein to Creatinine Ratio (UPCR) at Week 48
Description: Change from baseline in UPCR at Week 48 was reported.
Time Frame: Baseline and Week 48
Population: as for outcome 6
Measure: Median (Full Range); unit: milligram per gram (mg/g)
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch)
Number analyzed (Participants) | 336 | 325
milligram per gram (mg/g) | -15.72 (-748.1) [-748.1 to 254.2] | -10.53 (-903.0) [-903.0 to 1546.1]
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) vs DRV/COBI+ FTC/TDF (Control) (Baseline to Switch); Test type: Other; p = 0.033, Wilcoxon rank sum test

12. Secondary Outcome: Change From Baseline in Urine Albumin to Creatinine Ratio (UACR) at Week 48
Description: Change from baseline in UACR at Week 48 was reported.
Time Frame: Baseline and Week 48
Population: as for outcome 6
Measure: Median (Full Range); unit: mg/g
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch)
Number analyzed (Participants) | 338 | 327
mg/g | -0.58 (-226.5) [-226.5 to 143.8] | -0.15 (-640.4) [-640.4 to 969.6]
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) vs DRV/COBI+ FTC/TDF (Control) (Baseline to Switch); Test type: Other; p = 0.033, Wilcoxon rank sum test

13. Secondary Outcome: Change From Baseline in Urine Retinol Binding Protein To Creatinine Ratio (URBPCR) at Week 48
Description: Change from baseline in URBPCR at Week 48 were reported.
Time Frame: Baseline and Week 48
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Here, N (number of participant analyzed) signifies participants evaluated for this outcome measure.
Measure: Median (Full Range); unit: microgram per gram (mcg/g)
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch)
Number analyzed (Participants) | 334 | 324
microgram per gram (mcg/g) | 7.00 (-1555.7) [-1555.7 to 5183.8] | 35.02 (-700.7) [-700.7 to 30350.2]
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) vs DRV/COBI+ FTC/TDF (Control) (Baseline to Switch); Test type: Other; p < 0.001, Wilcoxon rank sum test

14. Secondary Outcome: Change From Baseline in Urine Beta-2 Microglobulin to Creatinine Ratio (UB2MGCR) at Week 48
Description: Change from baseline in UB2MGCR at Week 48 were reported.
Time Frame: Baseline and Week 48
Population: as for outcome 13
Measure: Median (Full Range); unit: mcg/g
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch)
Number analyzed (Participants) | 331 | 320
mcg/g | -30.42 (-11818.6) [-11818.6 to 3452.0] | 18.36 (-2440.5) [-2440.5 to 90832.0]
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) vs DRV/COBI+ FTC/TDF (Control) (Baseline to Switch); Test type: Other; p < 0.001, Wilcoxon rank sum test

15. Secondary Outcome: Percent Change From Baseline in Urine Fractional Excretion of Phosphate (FEPO4) at Week 48
Description: Percent change from baseline in FEPO4 at Week 48 was reported.
Time Frame: Baseline and Week 48
Population: as for outcome 6
Measure: Median (Full Range); unit: Percent change
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch)
Number analyzed (Participants) | 339 | 329
Percent change | 16.00 (-87.3) [-87.3 to 1756.6] | 22.55 (-90.1) [-90.1 to 1720.7]
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) vs DRV/COBI+ FTC/TDF (Control) (Baseline to Switch); Test type: Other; p = 0.147, Wilcoxon rank sum test

16. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time of Administration to 24 Hours Post-dose (AUC0-24h) of Darunavir
Description: AUC (0-24) is the area under the plasma concentration-time curve from time zero to 24 hours post-dose.
Time Frame: 0 to 24 hours post dose
Population: Pharmacokinetic (PK) analysis set included all participants who were randomized, received at least 1 dose of study drug and plasma concentration data for analytes of interest were available. PK data of DRV was analyzed only for test arm as per planned analyses. Here, 'N' (number of participants analyzed) number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours*nanogram per milliliter (h*ng/mL)
Groups:
- Darunavir 800 mg [D/C/F/TAF]: Participants received DRV 800 mg along with COBI 150 mg, FTC 200 mg, TAF 10 mg as a (D/C/F/TAF) FDC oral tablet once daily along with DRV/COBI FDC-matching placebo and FTC/TDF FDC-matching placebo tablets once daily up to Week 48.
Arm/Group | Darunavir 800 mg [D/C/F/TAF]
Number analyzed (Participants) | 355
hours*nanogram per milliliter (h*ng/mL) | 87909.3282 (20232.09905)

17. Secondary Outcome: Predose (Trough) Plasma Concentration (C0h) of Darunavir
Description: C0h is defined as the predose (trough) plasma concentration or concentration just prior to study drug administration.
Time Frame: 30 minutes to 4 hours postdose at Weeks 2, 4, 12, 24 and 48 and at 2 timepoints with at least 2.5 hours in between sampling at Week 8 and 36 (first sample between 1 and 4 hours postdose)
Population: PK analysis set included all participants who were randomized, received at least 1 dose of study drug and plasma concentration data for analytes of interest were available. PK data of DRV was analyzed only for test arm as per planned analyses. Here, 'N' (number of participants analyzed) number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Darunavir 800 mg [D/C/F/TAF (Test)]: Participants received DRV 800 mg along with COBI 150 mg, FTC 200 mg, TAF 10 mg as a (D/C/F/TAF) FDC oral tablet once daily along with DRV/COBI FDC-matching placebo and FTC/TDF FDC-matching placebo tablets once daily up to Week 48.
Arm/Group | Darunavir 800 mg [D/C/F/TAF (Test)]
Number analyzed (Participants) | 355
nanogram per milliliter (ng/mL) | 1898.9100 (758.83837)

18. Secondary Outcome: Area Under the Plasma Concentration Time Curve Across the Dosing Interval (AUCtau) of Tenofovir Alafenamide
Description: The AUCtau is the measure of the plasma drug concentration from time zero to end of dosing interval. It is used to characterize drug absorption.
Time Frame: as for outcome 17
Population: PK analysis set included all participants who were randomized, received at least 1 dose of study drug and plasma concentration data for analytes of interest were available. PK data of TAF was analyzed only for test arm as per planned analyses. Here, 'N' (number of participants analyzed) number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Tenofovir Alafenamide 10 mg [D/C/F/TAF (Test)]: Participants received TAF 10 mg along with DRV 800 mg, COBI 150 mg, FTC 200 mg as a (D/C/F/TAF) FDC oral tablet once daily along with DRV/COBI FDC-matching placebo and FTC/TDF FDC-matching placebo tablets once daily up to Week 48.
Arm/Group | Tenofovir Alafenamide 10 mg [D/C/F/TAF (Test)]
Number analyzed (Participants) | 355
h*ng/mL | 132.3117 (40.87742)

19. Secondary Outcome: Plasma Concentrations 2 Hours After Dosing (C0-2h) of Tenofovir Alafenamide
Description: C0-2h is defined as the plasma concentrations 2 hours after dosing.
Time Frame: 0 to 2 hours post dose
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tenofovir Alafenamide 10 mg [D/C/F/TAF (Test)]
Number analyzed (Participants) | 355
ng/mL | 11.9785 (11.86104)

20. Secondary Outcome: Percent Change From Baseline in Hip and Spine Bone Mineral Density (BMD)
Description: The BMD is the amount of mineral in gram per square centimeter of bone, which was assessed by dual energy x-ray absorptiometry (DEXA) scan. Positive values are "best values" and negative values are "worst values" of change. Percent change from baseline in hip and spine BMD was assessed.
Time Frame: Baseline, Weeks 24 and 48
Population: Bone investigation substudy (BIS) analysis set included all participants who were randomized, received at least 1 dose of study drug in study and had at least one post-baseline value for either biomarker/BMD data. Here, n (number analyzed) signifies participants analyzed for this OM at specified timepoints.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch)
Number analyzed (Participants) | 113 | 99
Percent change
  Hip region BMD (Week 24): number analyzed (Participants) | 97 | 82
  Hip region BMD (Week 24) | 0.29 (0.248) | -1.66 (0.269)
  Spine region BMD (Week 24): number analyzed (Participants) | 96 | 82
  Spine region BMD (Week 24) | -1.34 (0.285) | -3.43 (0.309)
  Hip region BMD (Week 48): number analyzed (Participants) | 96 | 85
  Hip region BMD (Week 48) | 0.17 (0.322) | -2.69 (0.342)
  Spine region BMD (Week 48): number analyzed (Participants) | 96 | 85
  Spine region BMD (Week 48) | -0.68 (0.402) | -2.38 (0.428)
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) vs DRV/COBI+ FTC/TDF (Control) (Baseline to Switch); Hip region BMD (Week 24); Test type: Other; p < 0.001, ANCOVA; LS mean difference = 1.95, 95% CI 2-sided [1.227 to 2.678], Standard Error of Mean 0.368
Statistical Analysis 2: Comparison: D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) vs DRV/COBI+ FTC/TDF (Control) (Baseline to Switch); Hip region BMD (Week 48); Test type: Other; p < 0.001, ANCOVA; LS mean difference = 2.86, 95% CI 2-sided [1.934 to 3.791], Standard Error of Mean 0.470
Statistical Analysis 3: Comparison: D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) vs DRV/COBI+ FTC/TDF (Control) (Baseline to Switch); Spine region BMD (Week 24); Test type: Other; p < 0.001, ANCOVA; LS mean difference = 2.09, 95% CI 2-sided [1.259 to 2.919], Standard Error of Mean 0.421
Statistical Analysis 4: Comparison: D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) vs DRV/COBI+ FTC/TDF (Control) (Baseline to Switch); Spine region BMD (Week 48); Test type: Other; p = 0.004, ANCOVA; LS mean difference = 1.70, 95% CI 2-sided [0.539 to 2.858], Standard Error of Mean 0.588

21. Secondary Outcome: Change From Baseline in BMD T-score of Hip and Spine
Description: BMD status was assessed using BMD T-scores; normal bone status was defined by a BMD T-score >= -1, osteopenia by a T-score >= -2.5 to <-1.0, and osteoporosis by a T-score <-2.5.
Time Frame: Baseline, Weeks 24 and 48
Population: BIS analysis set included all participants who were randomized, received at least 1 dose of study drug in study and had at least one post-baseline value for either biomarker/BMD data. Here, 'n' (number analyzed) signifies participants analyzed for this outcome measure at specified timepoints.
Measure: Mean (Standard Error); unit: BMD T-score
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch)
Number analyzed (Participants) | 113 | 99
BMD T-score
  Hip region BMD T-score (Week 24): number analyzed (Participants) | 97 | 82
  Hip region BMD T-score (Week 24) | 0.019 (0.0180) | -0.109 (0.0157)
  Spine region BMD T-score (Week 24): number analyzed (Participants) | 96 | 82
  Spine region BMD T-score (Week 24) | -0.121 (0.0259) | -0.322 (0.0307)
  Hip region BMD T-score (Week 48): number analyzed (Participants) | 96 | 85
  Hip region BMD T-score (Week 48) | 0.015 (0.0213) | -0.177 (0.0225)
  Spine region BMD T-score (Week 48): number analyzed (Participants) | 96 | 85
  Spine region BMD T-score (Week 48) | -0.061 (0.0390) | -0.225 (0.0386)

22. Secondary Outcome: Change From Baseline in Alkaline Phosphatase (ALP) Levels at Weeks 24 and 48
Description: Change from baseline in ALP at Weeks 24 and 48 was reported.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 21
Measure: Mean (Standard Error); unit: Units per liter (U/L)
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch)
Number analyzed (Participants) | 113 | 99
Units per liter (U/L)
  Week 24: number analyzed (Participants) | 103 | 88
  Week 24 | -3.2 (1.17) | 12.0 (1.74)
  Week 48: number analyzed (Participants) | 97 | 85
  Week 48 | -1.1 (1.29) | 15.1 (2.00)

23. Secondary Outcome: Change From Baseline in Levels of Serum Procollagen 1 N-Terminal Propeptide (P1NP) at Weeks 24 and 48
Description: Change from baseline in serum P1NP at Weeks 24 and 48 were reported.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 21
Measure: Mean (Standard Error); unit: microgram per liter (mcg/L)
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch)
Number analyzed (Participants) | 113 | 99
microgram per liter (mcg/L)
  Week 24: number analyzed (Participants) | 101 | 95
  Week 24 | 1.892 (1.3754) | 24.679 (2.0956)
  Week 48: number analyzed (Participants) | 96 | 84
  Week 48 | 0.065 (1.6428) | 24.251 (2.6337)

24. Secondary Outcome: Change From Baseline in Levels of Serum Collagen Type 1 Beta Carboxy Telopeptide (CTX) at Weeks 24 and 48
Description: Change from baseline in serum CTX at Weeks 24 and 48 were reported.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 21
Measure: Mean (Standard Error); unit: mcg/L
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch)
Number analyzed (Participants) | 113 | 99
mcg/L
  Week 24: number analyzed (Participants) | 103 | 83
  Week 24 | 0.047 (0.0165) | 0.283 (0.0251)
  Week 48: number analyzed (Participants) | 97 | 81
  Week 48 | 0.046 (0.0174) | 0.226 (0.0234)

25. Secondary Outcome: Change From Baseline in Levels of Parathyroid Hormone (PTH) at Weeks 24 and 48
Description: Change from baseline in PTH at Weeks 24 and 48 were reported.
Time Frame: Baseline, Weeks 24 and 48
Population: BIS analysis set included participants who were randomized, received at least 1 dose of study drug in study and had at least one post-baseline value for either biomarker/BMD data. Here, 'n' (number analyzed) signifies participants analyzed for this outcome measure at specified timepoints.
Measure: Mean (Standard Error); unit: Picomol per liter (pmol/L)
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch)
Number analyzed (Participants) | 113 | 99
Picomol per liter (pmol/L)
  Week 24: number analyzed (Participants) | 101 | 83
  Week 24 | 0.113 (0.2171) | 0.777 (0.2401)
  Week 48: number analyzed (Participants) | 95 | 83
  Week 48 | -0.004 (0.2232) | 0.633 (0.2155)

26. Secondary Outcome: Change From Baseline in Levels of 25-Hydroxyvitamin D (25-OH Vitamin D), at Week 24 and 48
Description: Change from baseline in 25-OH Vitamin D levels at Week 24 and 48 were reported.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 21
Measure: Mean (Standard Error); unit: nanomol per liter (nmol/L)
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch)
Number analyzed (Participants) | 113 | 99
nanomol per liter (nmol/L)
  Week 24: number analyzed (Participants) | 101 | 84
  Week 24 | 12.7 (2.76) | 22.1 (3.76)
  Week 48: number analyzed (Participants) | 97 | 82
  Week 48 | 16.9 (2.84) | 28.3 (3.15)

27. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies Per mL at Week 96 Defined by FDA Snapshot Approach
Description: Percentage of participants with a HIV-1 RNA < 50 copies per mL were assessed using FDA snapshot approach which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status. The snapshot approach classified participants into 3 outcome categories: 1) virologic success (HIV RNA < 20/50/200 copies per mL at Week 96), 2) virologic failure (HIV RNA greater than or equal to [>=] 20/50/200 copies per mL at Week 96), 3) no viral load data in the Week 96 visit window (discontinued due to adverse event/death/other reason). The missing HIV-1 RNA is considered as non-response.
Time Frame: At Week 96
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 362 | 291
percentage of participants | 85.1 (81.0) [81.0 to 88.6] | 94.2 (90.8) [90.8 to 96.6]

28. Secondary Outcome: Change From Reference in log10 HIV-1 RNA Levels at Week 96
Description: Change from reference in log10 HIV-1 RNA levels were reported. Here, reference 1 is the comparative phase baseline value in Week 48 analysis for Test group and reference 2 is the last value prior to the switch for Control group.
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Based on not completed (NC) equal to (=) failure (F) analysis with values after discontinuation imputed with the baseline value. Other (intermittent) missing values are imputed using last observation carried forward (LOCF). Here N (number of participants analyzed) signifies participants evaluated for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: log10 HIV-1 RNA copies per mL
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 362 | 289
log10 HIV-1 RNA copies per mL | -2.72 (0.0614) | -0.0027 (0.0131)

29. Secondary Outcome: Change From Reference in CD4+ Cell Count at Week 96
Description: The immunologic change was determined by changes in cluster of differentiation (CD4+) cell count. Change from reference in CD4+ cell count at Week 96 was assessed. Here, reference 1 is the comparative phase baseline value in Week 48 analysis for test group and reference 2 is the last value prior to the switch for Control group.
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Based on NC=F analysis with values after discontinuation imputed with the baseline value. Other (intermittent) missing values are imputed using LOCF. Here, N (number of participants analyzed) signifies participants evaluated for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: cells/mm^3
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 362 | 289
cells/mm^3 | 228.85 (11.951) [lower limit 11.951] | 27.01 (9.522) [lower limit 9.522]

30. Secondary Outcome: Percentage of Participants With >95% Treatment Adherence Assessed by Drug Accountability
Description: Treatment adherence assessed by drug accountability (based on pill count) from start of treatment/switch to last study drug intake by determination of the cumulative treatment adherence in participants who returned all dispensed bottles prior to or at the last visit in the study. Adherent participants were defined as having an adherence >95% as assessed by drug accountability.
Time Frame: Baseline to Switch and switch to EOE to Open-Label D/C/F/TAF (Up to 3 years)
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Here, N (number of participants analyzed) signifies participants evaluated for this outcome measure and n (number analyzed) signifies participants analyzed for this outcome measure at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch) | Switch to D/C/F/TAF
Number analyzed (Participants) | 289 | 282 | 222
percentage of participants
  Baseline to Switch (double-blind treatment): number analyzed (Participants) | 289 | 282 | 0
  Baseline to Switch (double-blind treatment) | 87.2 | 82.6 |
  Switch to End of Extension (open-label D/C/F/TAF): number analyzed (Participants) | 231 | 0 | 222
  Switch to End of Extension (open-label D/C/F/TAF) | 92.2 |  | 88.7

31. Secondary Outcome: Percentage of Participants With Grade 3 and 4 Adverse Events (AEs), Serious Adverse Events (SAEs), and Premature Discontinuations Due to Adverse Events Through Week 96
Description: as for outcome 10
Time Frame: Up to Week 96
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. This outcome measure was planned to be reported for participants who received D/C/F/TAF in group 1 and who switched to D/C/F/TAF in group 2.
Measure: Number; unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 362 | 295
percentage of participants
  Grade 3 AEs | 11.6 | 3.7
  Grade 4 AEs | 0.8 | 1.4
  SAEs | 10.8 | 2.7
  Premature discontinuations due to AEs | 2.8 | 0.3

32. Secondary Outcome: Change From Reference in Serum Creatinine
Description: Change from reference in serum creatinine was reported. Here, reference 1 is the comparative phase baseline value in Week 48 analysis for test group and reference 2 is the last value prior to the switch for Control group.
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Here, N (number of participants analyzed) signifies participants evaluated for this outcome measure. This outcome measure was planned to be reported for participants who received D/C/F/TAF in Test group and who switched to D/C/F/TAF in Switch to D/C/F/TAF group.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 317 | 287
mg/dL | 0.045 (-0.25) [-0.25 to 0.30] | -0.034 (-0.71) [-0.71 to 0.40]

33. Secondary Outcome: Change From Reference in eGFRcr by CKD-EPI Formula
Description: Change from reference in eGFRcr was calculated using the CKD-EPI equation as per Stage 1 (normal or high GFR) to Stage 5 (End Stage of CKD). The eGFRcr was assessed by calculating serum creatinine (Scr) using the CKD-EPI equation: eGFRcr milliliter per minute per 1.72 meter square (mL/min/1.73m^2) = 144 * (Scr/0.7)^-0.329 * 0.993^age (Scr =< 0.7 mg/dL) and eGFRcr mL/min/1.73m^2 = 144 * (Scr/0.7)^-1.209 * 0.993^age (Scr >0.7 mg/dL) for female participants and eGFRcr mL/min/1.73m^2 = 141 x (Scr/0.9)^-0.411 x 0.993^age (Scr =<0.9 mg/dL) and eGFRcr mL/min/1.73m^2 = 141 * (Scr/0.9)^-1.209 x 0.993^age (Scr >0.9 mg/dL) for male participants. Here, reference 1 is the comparative phase baseline value in Week 48 analysis for test group and reference 2 is the last value prior to the switch for Control group.
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: as for outcome 32
Measure: Median (Full Range); unit: mL/min/1.73 m^2
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 317 | 287
mL/min/1.73 m^2 | -5.6 (-33) [-33 to 29] | 2.3 (-29) [-29 to 43]

34. Secondary Outcome: Change From Reference in Estimated Glomerular Filtration Rate Based on Serum Creatinine by Cockcroft-Gault Formula
Description: Change from reference in eGFRcr by cockcroft-gault formula was reported. The eGFRcr was assessed by calculated creatinine clearance (CrCl) using the Cockcroft-Gault formula, and was assessed using CrCl [mL/min] = (140 - A) * W / (72 * C) * R. Where A is age at sample date [years], W is body weight at specific visit (kilogram [kg]), C is the serum concentration of creatinine [mg/dL], R = 1 if the participant is male and = 0.85 if female. Here, reference 1 is the comparative phase baseline value in Week 48 analysis for test group and reference 2 is the last value prior to the switch for Control group.
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: as for outcome 32
Measure: Median (Full Range); unit: mL/min
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 317 | 287
mL/min | -5.2 (-73) [-73 to 41] | 4.6 (-47) [-47 to 55]

35. Secondary Outcome: Change From Reference in Estimated Glomerular Filtration Rate Based on Serum Cystatin C (eGFRcyst) by CKD-EPI Formula
Description: Change from reference in eGFRcyst was calculated using the CKD-EPI equation as per Stage 1 (normal or high GFR) to Stage 5 (End Stage of CKD): <15 mL/min indicate very severe or end stage kidney failure. The eGFRcyst was assessed by calculated serum cystatin C (Scyst) using the CKD-EPI equation: eGFRcyst mL/min/1.73m^2 = 133 * (Scyst/0,8)^-0.499 * 0.996^age [x 0.932 if female] (Scyst =<0.8 mg/L) and eGFRcr mL/min/1.73m^2 = 133 * (Scyst/0,8)^-1.328 * 0.996^age [* 0.932 if male] (Scyst >0.8 mg/L). Here, reference 1 is the comparative phase baseline value in Week 48 analysis for test group and reference 2 is the last value prior to the switch for Control group.
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: as for outcome 32
Measure: Median (Full Range); unit: mL/min/1.73 m^2
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 22 | 33
mL/min/1.73 m^2 | 4.4 (-14) [-14 to 37] | 0 (-12) [-12 to 26]

36. Secondary Outcome: Change From Reference in UPCR
Description: Change from reference in UPCR was reported. Here, reference 1 is the comparative phase baseline value in Week 48 analysis for test group and reference 2 is the last value prior to the switch for Control group.
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF+ FTC/TDF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: as for outcome 32
Measure: Median (Full Range); unit: mg/g
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 312 | 282
mg/g | -15.46 [-728.7 to 197.9] | -1.40 [-705.7 to 289.2]

37. Secondary Outcome: Change From Reference in UACR
Description: Change from reference in UACR at Week 96 was reported. Here, reference 1 is the comparative phase baseline value in Week 48 analysis for test group and reference 2 is the last value prior to the switch for Control group.
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: as for outcome 32
Measure: Median (Full Range); unit: mg/g
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 317 | 287
mg/g | -0.70 (-288.1) [-288.1 to 44.5] | -0.49 (-294.5) [-294.5 to 583.2]

38. Secondary Outcome: Change From Reference in URBPCR
Description: Change from reference in URBPCR at Week 96 were reported. Here, reference 1 is the comparative phase baseline value in Week 48 analysis for test group and reference 2 is the last value prior to the switch for Control group.
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: as for outcome 32
Measure: Median (Full Range); unit: mcg/g
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 313 | 285
mcg/g | 13.70 (-1555.1) [-1555.1 to 2547.1] | -35.53 (-108886.3) [-108886.3 to 291.3]

39. Secondary Outcome: Change From Reference in UB2MGCR
Description: Change from reference in UB2MGCR was reported. Here, reference 1 is the comparative phase baseline value in Week 48 analysis for test group and reference 2 is the last value prior to the switch for Control group.
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: as for outcome 32
Measure: Median (Full Range); unit: mcg/g
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 310 | 286
mcg/g | -27.04 (-11704.6) [-11704.6 to 894.7] | -40.53 (-111778.9) [-111778.9 to 624.6]

40. Secondary Outcome: Percent Change From Reference in Urine FEPO4
Description: Percent change from reference in FEPO4 at Week 96 were reported. Here, reference 1 is the comparative phase baseline value in Week 48 analysis for test group and reference 2 is the last value prior to the switch for Control group.
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Here, 'N' (number of participants analyzed) signifies participants evaluated for this outcome measure. This outcome measure was planned to be reported for participants who received D/C/F/TAF in Test group and who switched to D/C/F/TAF in Switch to D/C/F/TAF group.
Measure: Median (Full Range); unit: Percent change in urine FEPO4
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 316 | 286
Percent change in urine FEPO4 | 18.52 (-84.2) [-84.2 to 1170.1] | -7.51 (-83.5) [-83.5 to 494.7]

41. Secondary Outcome: Percent Change From Reference in Hip and Spine BMD
Description: The BMD is the amount of mineral in gram per square centimeter of bone, which was assessed by DEXA scan. Positive values are "best values" and negative values are "worst values" of change. Percent change from reference in hip and spine BMD was assessed. Here, reference 1 is the comparative phase baseline value in Week 48 analysis for test group and reference 2 is the last value prior to the switch for Control group.
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: The analysis population is BIS. Here, 'N' (number of participants analyzed) signifies participants evaluated for this outcome measure and 'n' (number analyzed) signifies participants analyzed for this outcome measure at specified category. This outcome measure was planned to be reported for participants who received D/C/F/TAF in Test group and who switched to D/C/F/TAF in Switch to D/C/F/TAF group.
Measure: Mean (Standard Error); unit: Percent change in BMD
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 113 | 83
Percent change in BMD
  Hip region BMD: number analyzed (Participants) | 87 | 71
  Hip region BMD | -0.2565 (0.35599) | 0.5467 (0.38512)
  Spine region BMD: number analyzed (Participants) | 86 | 71
  Spine region BMD | -0.9349 (0.44599) | 0.4829 (0.39270)

42. Secondary Outcome: Change From Reference in BMD T-score of Hip and Spine at Week 96
Description: BMD status was assessed using BMD T-scores; normal bone status was defined by a BMD T-score >= -1, osteopenia by a T-score >= -2.5 to <-1.0, and osteoporosis by a T-score <-2.5. Here, reference 1 is the comparative phase baseline value in Week 48 analysis for test group and reference 2 is the last value prior to the switch for Control group.
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: The analysis set of BIS. Here, 'N' (number of participants analyzed) signifies participants evaluated for this outcome measure and n (number analyzed) signifies participants analyzed for this endpoint at specified category. This outcome measure was planned to be reported for participants who received D/C/F/TAF in Test group and who switched to D/C/F/TAF in Switch to D/C/F/TAF group.
Measure: Mean (Standard Error); unit: BMD T-score
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 87 | 71
BMD T-score
  Hip region BMD T-score | -0.016 (0.0245) | 0.025 (0.0272)
  Spine region BMD T-score: number analyzed (Participants) | 86 | 71
  Spine region BMD T-score | -0.090 (0.0407) | 0.034 (0.0355)

43. Secondary Outcome: Change From Reference in ALP Levels
Description: Change from reference in ALP levels at Week 96 was reported. Here, reference 1 is the comparative phase baseline value in Week 48 analysis for test group and reference 2 is the last value prior to the switch for Control group.
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: The analysis population is BIS. Here, N (number of participants analyzed) signifies participants evaluated for this outcome measure. This outcome measure was planned to be reported for participants who received D/C/F/TAF in Test group and who switched to D/C/F/TAF in Switch to D/C/F/TAF group.
Measure: Mean (Standard Error); unit: U/L
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 92 | 80
U/L | -0.9 (1.23) [lower limit 1.23] | -9.7 (1.55) [lower limit 1.55]

44. Secondary Outcome: Change From Reference in Levels of Serum P1NP
Description: Change from reference in serum P1NP levels were reported. Here, reference 1 is the comparative phase baseline value in Week 48 analysis for test group and reference 2 is the last value prior to the switch for Control group.
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: BIS analysis set included all participants who were randomized, received at least 1 dose of study drug in study and had at least one post-baseline value for either biomarker/BMD data. Here, N (number of participants analyzed) signifies participants evaluated for this outcome measure. This outcome measure was planned to be reported for participants who received D/C/F/TAF in Test group and who switched to D/C/F/TAF in Switch to D/C/F/TAF group.
Measure: Mean (Standard Error); unit: mcg/L
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 91 | 75
mcg/L | 2.817 (1.7140) | -11.963 (1.7636)

45. Secondary Outcome: Change From Reference in Levels of Serum CTX
Description: Change from reference in serum CTX levels were reported. Here, reference 1 is the comparative phase baseline value in Week 48 analysis for test group and reference 2 is the last value prior to the switch for Control group.
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: as for outcome 44
Measure: Mean (Standard Error); unit: mcg/L
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 91 | 77
mcg/L | 0.041 (0.0190) [lower limit 0.0190] | -0.162 (0.0190) [lower limit 0.0190]

46. Secondary Outcome: Change From Reference in Levels of PTH
Description: Change from reference in PTH levels were reported. Here, reference 1 is the comparative phase baseline value in Week 48 analysis for test group and reference 2 is the last value prior to the switch for Control group.
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: as for outcome 44
Measure: Mean (Standard Error); unit: pmol/L
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 90 | 77
pmol/L | -0.290 (0.2078) [lower limit 0.2078] | -1.283 (0.2483) [lower limit 0.2483]

47. Secondary Outcome: Change From Reference in Levels of 25-OH Vitamin D
Description: Change from reference in 25-OH Vitamin D were reported. Here, reference 1 is the comparative phase baseline value in Week 48 analysis for test group and reference 2 is the last value prior to the switch for Control group.
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: as for outcome 44
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 91 | 77
nmol/L | 21.3 (2.45) [lower limit 2.45] | -10.3 (2.87) [lower limit 2.87]

48. Secondary Outcome: Percentage of Participants With HIV RNA <50, <20, and <200 Copies/mL Post-week 96 to End of Extension
Description: Percentage of participants with HIV RNA <50, <20, and <200 copies/mL post Week 96 to end of extension were reported.
Time Frame: Week 96 to end of extension (up to 3 years)
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Here, 'N' (number of participants analyzed) signifies participants evaluated for this outcome measure and n (number analyzed) signifies participants analyzed for this outcome measure at specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 303 | 296
percentage of participants
  Week 96 + 6 months (<50 copies/mL) | 97.7 [95.3 to 99.1] | 96.3 [93.4 to 98.1]
  Week 96 + 12 months (<50 copies/mL): number analyzed (Participants) | 194 | 214
  Week 96 + 12 months (<50 copies/mL) | 99.0 [96.3 to 99.9] | 96.7 [93.4 to 98.7]
  Week 96 + 18 months (<50 copies/mL): number analyzed (Participants) | 158 | 167
  Week 96 + 18 months (<50 copies/mL) | 98.1 [94.6 to 99.6] | 98.2 [94.8 to 99.6]
  Week 96 + 24 months (<50 copies/mL): number analyzed (Participants) | 81 | 92
  Week 96 + 24 months (<50 copies/mL) | 97.5 [91.4 to 99.7] | 95.7 [89.2 to 98.8]
  Week 96 + 30 months (<50 copies/mL): number analyzed (Participants) | 57 | 58
  Week 96 + 30 months (<50 copies/mL) | 94.7 [85.4 to 98.9] | 91.4 [81.0 to 97.1]
  Week 96 + 36 months (<50 copies/mL): number analyzed (Participants) | 19 | 16
  Week 96 + 36 months (<50 copies/mL) | 100.0 [82.4 to 100.0] | 68.8 [41.3 to 89.0]
  Week 96 + 6 months (<20 copies/mL) | 85.8 [81.4 to 89.5] | 88.2 [83.9 to 91.6]
  Week 96 + 12 months (<20 copies/mL): number analyzed (Participants) | 194 | 214
  Week 96 + 12 months (<20 copies/mL) | 89.7 [84.5 to 93.6] | 91.6 [87.0 to 94.9]
  Week 96 + 18 months (<20 copies/mL): number analyzed (Participants) | 158 | 167
  Week 96 + 18 months (<20 copies/mL) | 92.4 [87.1 to 96.0] | 92.8 [87.8 to 96.2]
  Week 96 + 24 months (<20 copies/mL): number analyzed (Participants) | 81 | 92
  Week 96 + 24 months (<20 copies/mL) | 90.1 [81.5 to 95.6] | 87.0 [78.3 to 93.1]
  Week 96 + 30 months (<20 copies/mL): number analyzed (Participants) | 57 | 58
  Week 96 + 30 months (<20 copies/mL) | 89.5 [78.5 to 96.0] | 84.5 [72.6 to 92.7]
  Week 96 + 36 months (<20 copies/mL): number analyzed (Participants) | 19 | 16
  Week 96 + 36 months (<20 copies/mL) | 94.7 [74.0 to 99.9] | 62.5 [35.4 to 84.8]
  Week 96 + 6 months (<200 copies/mL) | 99.7 [98.2 to 100.0] | 99.3 [97.6 to 99.9]
  Week 96 + 12 months (<200 copies/mL): number analyzed (Participants) | 194 | 214
  Week 96 + 12 months (<200 copies/mL) | 100.0 [98.1 to 100.0] | 99.5 [97.4 to 100]
  Week 96 + 18 months (<200 copies/mL): number analyzed (Participants) | 158 | 167
  Week 96 + 18 months (<200 copies/mL) | 98.7 [95.5 to 99.8] | 98.2 [94.8 to 99.6]
  Week 96 + 24 months (<200 copies/mL): number analyzed (Participants) | 81 | 92
  Week 96 + 24 months (<200 copies/mL) | 97.5 [91.4 to 99.7] | 97.8 [92.4 to 99.7]
  Week 96 + 30 months (<200 copies/mL): number analyzed (Participants) | 57 | 58
  Week 96 + 30 months (<200 copies/mL) | 96.5 [87.9 to 99.6] | 98.3 [90.8 to 100.0]
  Week 96 + 36 months (<200 copies/mL): number analyzed (Participants) | 19 | 16
  Week 96 + 36 months (<200 copies/mL) | 100.0 [82.4 to 100.0] | 87.5 [61.7 to 98.4]

49. Secondary Outcome: Percentage of Participants With Protocol-defined Virologic Failure (PDVF)
Description: Percentage of participants with PDVF were reported. Protocol-defined virologic failure was defined as having virologic non-response (HIV-1 RNA <1 log10 reduction from baseline and >=50 copies/mL at the Week 8 visit, confirmed at the next visit), virologic rebound (confirmed HIV-1 RNA >=50 copies/mL after confirmed consecutive HIV-1 RNA <50 copies/mL or confirmed >1 log10 increase in HIV-1 RNA from nadir), or viremic at final time point (final available on treatment HIV-1 RNA >=400 copies/mL).
Time Frame: From Baseline up to Week 96
Population: The analysis population is ITT. Here, n (number analyzed) signifies participants analyzed for this OM at specified timepoints. Participants received treatment from baseline till Week 48/Switch in control arm and from switch till Week 96 in Switch to D/C/F/TAF arm. Therefore, Week 96 and Week 48 data was not collected for both arms at respective timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch) | Switch to D/C/F/TAF
Number analyzed (Participants) | 362 | 363 | 295
percentage of participants
  Participants who met PDVF (Baseline - Week 96): number analyzed (Participants) | 362 | 0 | 0
  Participants who met PDVF (Baseline - Week 96) | 4.1 |  |
  Virologic non-response (Baseline - Week 96): number analyzed (Participants) | 362 | 0 | 0
  Virologic non-response (Baseline - Week 96) | 0.6 |  |
  Virologic rebound (Baseline-Week 96): number analyzed (Participants) | 362 | 0 | 0
  Virologic rebound (Baseline-Week 96) | 0.3 |  |
  Viremic at final time point (Baseline-Week 96): number analyzed (Participants) | 362 | 0 | 0
  Viremic at final time point (Baseline-Week 96) | 0.6 |  |
  Participants who met PDVF (Baseline - Switch): number analyzed (Participants) | 0 | 363 | 0
  Participants who met PDVF (Baseline - Switch) |  | 4.4 |
  Virologic non-response (Baseline - Switch): number analyzed (Participants) | 0 | 363 | 0
  Virologic non-response (Baseline - Switch) |  | 0 |
  Virologic rebound (Baseline - Switch): number analyzed (Participants) | 0 | 363 | 0
  Virologic rebound (Baseline - Switch) |  | 3.9 |
  Viremic at final time point (Baseline - Switch): number analyzed (Participants) | 0 | 363 | 0
  Viremic at final time point (Baseline - Switch) |  | 0.6 |
  Participants who met PDVF (Switch - Week 96): number analyzed (Participants) | 0 | 0 | 295
  Participants who met PDVF (Switch - Week 96) |  |  | 1.1
  Virologic non-response (Switch - Week 96): number analyzed (Participants) | 0 | 0 | 295
  Virologic non-response (Switch - Week 96) |  |  | 0
  Virologic rebound (Switch - Week 96): number analyzed (Participants) | 0 | 0 | 295
  Virologic rebound (Switch - Week 96) |  |  | 1.1
  Viremic at final time point (Switch - Week 96): number analyzed (Participants) | 0 | 0 | 295
  Viremic at final time point (Switch - Week 96) |  |  | 0

50. Secondary Outcome: Percentage of Participants With PDVF Post-week 96 to End of Extension
Description: as for outcome 49
Time Frame: Week 96 to end of extension (up to 3 years)
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Here N (number of participants analyzed) refers to 311 for test group and 310 for switch to D/C/F/TAFgroup in below table.
Measure: Number; unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 311 | 310
percentage of participants
  Participants who met PDVF | 1.0 | 2.1
  Virologic non-response | 0 | 0
  Virologic rebound | 1.0 | 1.4
  Viremic at final time point | 0 | 0.7

51. Secondary Outcome: Percentage of Participants With Non-PDVF by Kaplan-Meier Estimates
Description: Percentage of participants with non-PDVF by Kaplan-Meier Estimates were reported. PDVF was defined as having virologic non-response (HIV-1 RNA <1 log10 reduction from baseline and >=50 copies/mL at the Week 8 visit, confirmed at the next visit), virologic rebound (confirmed HIV-1 RNA >=50 copies/mL after confirmed consecutive HIV-1 RNA <50 copies/mL or confirmed >1 log10 increase in HIV-1 RNA from nadir), or viremic at final time point (final available on treatment HIV-1 RNA >=400 copies/mL).
Time Frame: From Week 96 to end of extension (up to 2 years and 6 months)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 311 | 310
percentage of participants
  Week 96 | 100 [100 to 100] | 100 [100 to 100]
  Week 96 + 6 months | 99.6 [97.2 to 99.9] | 99.2 [97.0 to 99.8]
  Week 96 + 12 months | 99.6 [97.2 to 99.9] | 99.2 [97.0 to 99.8]
  Week 96 + 18 months | 98.6 [94.0 to 99.7] | 97.8 [94.1 to 99.2]
  Week 96 + 24 months | 97.3 [91.0 to 99.2] | 97.8 [94.1 to 99.2]
  Week 96 + 30 months | 97.3 [91.0 to 99.2] | 92.5 [79.8 to 97.3]

52. Secondary Outcome: Percentage of Participants With Time to Treatment Failure by Kaplan-Meier Estimates
Description: Percentage of participants with time to treatment failure by Kaplan-Meier Estimates were reported. Treatment failure was defined as having either protocol-defined virologic failure or having discontinued for reasons other than alternate access to D/C/F/TAF (or other ARVs).
Time Frame: From Week 96 to end of extension (up to 3 years)
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Here, n (number analyzed) signifies participants analyzed for this OM at specified timepoints.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 311 | 310
percentage of participants
  Week 96 | 100 [100 to 100] | 100 [100 to 100]
  Week 96 + 6 months | 98.9 [96.5 to 99.6] | 97.4 [94.5 to 98.7]
  Week 96 + 12 months | 95.6 [91.7 to 97.7] | 94.1 [90.2 to 96.5]
  Week 96 + 18 months | 90.6 [84.9 to 94.2] | 89.5 [84.3 to 93.0]
  Week 96 + 24 months | 87.1 [79.8 to 91.8] | 86.4 [80.0 to 90.9]
  Week 96 + 30 months | 84.8 [75.8 to 90.6] | 79.1 [68.9 to 86.3]
  Week 96 + 36 months: number analyzed (Participants) | 311 | 0
  Week 96 + 36 months | 84.8 [75.8 to 90.6] |

53. Secondary Outcome: CD4+ Cell Count Post-Week From 96 to End of Extension
Description: The immunologic change was determined by Cluster of CD4+ cell count. CD4+ cell count post-Week 96 to end of extension were assessed.
Time Frame: Week 96 to end of extension (up to 3 years)
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Here, N (number of participants analyzed) signifies participants evaluated for this outcome measure and n (number analyzed) signifies participants analyzed for this outcome measure at specified category.
Measure: Mean (Standard Error); unit: cells/mm^3
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 300 | 293
cells/mm^3
  Week 96 + 6 months | 790.2 (17.23) | 749.7 (16.44)
  Week 96 + 12 months: number analyzed (Participants) | 192 | 212
  Week 96 + 12 months | 779.4 (22.45) | 774.3 (21.91)
  Week 96 + 18 months: number analyzed (Participants) | 154 | 165
  Week 96 + 18 months | 789.8 (23.43) | 758.4 (23.25)
  Week 96 + 24 months: number analyzed (Participants) | 78 | 92
  Week 96 + 24 months | 781.9 (37.77) | 784.1 (30.78)
  Week 96 + 30 months: number analyzed (Participants) | 57 | 58
  Week 96 + 30 months | 741.6 (37.12) | 736.7 (37.47)
  Week 96 + 36 months: number analyzed (Participants) | 18 | 16
  Week 96 + 36 months | 784.7 (69.74) | 778.4 (86.59)

54. Secondary Outcome: Number of Participants With ARV Resistance
Description: Number of participants with DRV, FTC, TDF/TAF resistance were reported.
Time Frame: Baseline to end of extension (up to 4 years)
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Here, N (number of participants analyzed) signifies total number of participants with screening/baseline and endpoint genotype.
Measure: Count of Participants; unit: Participants
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch) | Switch to D/C/F/TAF
Number analyzed (Participants) | 12 | 8 | 7
Participants
  DRV resistance-associated mutations (RAMs) | 0 | 0 | 0
  TFV RAMs | 0 | 0 | 0
  FTC RAMs | 2 | 1 | 2

55. Secondary Outcome: Percentage of Participants With Grade 3 and 4 AEs, SAEs, and Premature Discontinuations Due to Adverse Events Post-Week 96 to End of Extension
Description: as for outcome 10
Time Frame: From Week 96 to end of extension (up to 3 years)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 311 | 310
percentage of participants
  Grade 3 AEs | 3.5 | 5.2
  Grade 4 AEs | 0 | 1.3
  SAEs | 3.2 | 4.8
  Premature discontinuations due to AEs | 1.0 | 1.3

ADVERSE EVENTS:
Time Frame: Up to 60 months
Description: The intent-to-treat (ITT) analysis set included all the participants who were randomized and received at least one dose of study treatment in the study.
Groups:
- D/C/F/TAF+ FTC/TDF (Test): Participants received a single oral tablet containing darunavir (DRV) 800 milligram (mg)/ cobicistat (COBI) 150 mg/ emtricitabine (FTC) 200 mg/ tenofovir alafenamide (TAF) 10 mg (D/C/F/TAF fixed dose combination [FDC]) once daily along with DRV/COBI FDC-matching placebo and FTC/tenofovir disoproxil fumarate (TDF) FDC-matching placebo tablets once daily up to Week 48 analysis unblinding visit (that is, after last participant has reached Week 48). After Week 48 analysis unblinding visit, all participants received D/C/F/TAF treatment up to Week 96 during the open-label, single-group treatment phase. After Week 96, participants were given the opportunity to continue D/C/F/TAF treatment during an extension phase until the D/C/F/TAF FDC tablet became commercially available.
- Switch to D/C/F/TAF Group: After Week 48 analysis unblinding visit, participants earlier receiving treatment with DRV/COBI+ FTC/TDF (Control) switched to D/C/F/TAF treatment and continued for up to Week 96 during open-label, single-group treatment phase. After Week 96, participants were given the opportunity to continue D/C/F/TAF treatment until the D/C/F/TAF FDC tablet became commercially available.
Arm/Group | D/C/F/TAF+ FTC/TDF (Test) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch) | Switch to D/C/F/TAF Group
All-Cause Mortality (participants affected / at risk) | 0/362 | 1/363 | 1/322
Serious Adverse Events (participants affected / at risk) | 47/362 | 36/363 | 21/322
Other Adverse Events (participants affected / at risk) | 284/362 | 252/363 | 137/322
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D/C/F/TAF+ FTC/TDF (Test) (N=362) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch) (N=363) | Switch to D/C/F/TAF Group (N=322)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Bone Marrow Oedema (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Anal Fistula (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Anogenital Dysplasia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza Like Illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Vascular Stent Stenosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis Sclerosing (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Abscess Limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anal Abscess (Infections and infestations) | 2 (3) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 3 (3) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea Infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis A (Infections and infestations) | 3 (3) | 3 (3) | 2 (2)
Hepatitis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Latent Syphilis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis Bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mumps (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Myocarditis Infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Neurosyphilis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Papilloma Viral Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Rectal Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Secondary Syphilis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Syphilis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Urethritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Exposure During Pregnancy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Intentional Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tendon Rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Waist Circumference Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Anogenital Warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 2 (2) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Kaposi's Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Squamous Cell Carcinoma of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness Postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Borderline Personality Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Drug Dependence (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1)
Calculus Urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Testicular Torsion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine Polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Toxic Skin Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Alcohol Use (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D/C/F/TAF+ FTC/TDF (Test) (N=362) | DRV/COBI+ FTC/TDF (Control) (Baseline to Switch) (N=363) | Switch to D/C/F/TAF Group (N=322)
Nasopharyngitis (Infections and infestations) | 64 (102) | 38 (58) | 19 (23)
Pharyngitis (Infections and infestations) | 31 (34) | 19 (24) | 7 (7)
Respiratory Tract Infection (Infections and infestations) | 20 (28) | 14 (22) | 8 (11)
Syphilis (Infections and infestations) | 41 (51) | 25 (29) | 24 (27)
Upper Respiratory Tract Infection (Infections and infestations) | 40 (55) | 30 (42) | 26 (43)
Diarrhoea (Gastrointestinal disorders) | 89 (143) | 72 (91) | 18 (20)
Nausea (Gastrointestinal disorders) | 34 (39) | 46 (56) | 8 (8)
Asthenia (General disorders) | 21 (21) | 15 (16) | 4 (4)
Fatigue (General disorders) | 26 (29) | 21 (24) | 1 (1)
Pyrexia (General disorders) | 20 (22) | 24 (28) | 6 (6)
Bronchitis (Infections and infestations) | 24 (32) | 25 (30) | 20 (22)
Chlamydial Infection (Infections and infestations) | 23 (27) | 9 (9) | 2 (2)
Gastroenteritis (Infections and infestations) | 28 (32) | 15 (15) | 5 (5)
Gonorrhoea (Infections and infestations) | 21 (31) | 14 (15) | 5 (6)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 28 (32) | 16 (16) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (25) | 17 (20) | 11 (12)
Back Pain (Musculoskeletal and connective tissue disorders) | 31 (36) | 10 (11) | 16 (18)
Osteopenia (Musculoskeletal and connective tissue disorders) | 19 (20) | 29 (32) | 0 (0)
Headache (Nervous system disorders) | 56 (79) | 38 (66) | 11 (12)
Anxiety (Psychiatric disorders) | 19 (21) | 9 (10) | 5 (5)
Insomnia (Psychiatric disorders) | 20 (24) | 13 (14) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (24) | 15 (16) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 37 (44) | 25 (26) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT02431247/Prot_002.pdf
  • Statistical Analysis Plan (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT02431247/SAP_003.pdf